CLINICAL TRIAL: NCT01473017
Title: Improving Mental Health in Diabetes: A Guided Self-Help Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11/NHS/0055
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2011-11

CONDITIONS: Type 2 Diabetes; Anxiety; Depression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT-based guided self-help (Experimental): Providing a guided self-help booklet to patients with anxiety/depression meeting criteria, with two telephone calls by a clinician to provide support with this.
  Interventions: Behavioral: CBT-based Guided Self-Help
- No CBT intervention (No Intervention): Control group in comparison to CBT guided self-help group

INTERVENTIONS:
Behavioral: CBT-based Guided Self-Help — CBT-based booklet tailored to anxiety and/or depression in Type 2 Diabetes to enhance mood and Diabetes self-care
  Arms: CBT-based guided self-help

SUMMARY:
This study employs a Randomised Controlled Trial design to investigate whether a CBT-based guided self-help intervention can improve anxiety, depression, psychological well-being, quality of life, Diabetic self-care and adherence; as compared to controls. The study aims to recruit 42 individuals with Diabetes and mild to moderate anxiety or depression. Anxiety and depression are common in patients with Type 2 Diabetes, and has been shown to affect Diabetes control. Literature suggests that CBT can benefit individuals with Diabetes and comorbid mental ill-health, however little research has been done to date on the effect of guided self-help in this population. It is expected that this intervention will improve patient's mental health, as well as extend the limited knowledge-base on guided self-help in chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of Type 2 Diabetes with mild-moderate anxiety and/or depression (scoring 8 to 15 on the HADS scale) will be recruited, provided they do not meet any one of the exclusion criteria listed below. Patients will be able to provide written informed consent.

Exclusion Criteria:

* Individuals with a history of clinically diagnosed psychotic symptoms, schizophrenia or bipolar disorder.
* Participants with a known Learning Disability or severe visual impairment.
* Participants who cannot read or write
* Participants under 18 years of age or over age 75
* Long-term hospital inpatients
* Individuals with a diagnosis of Diabetes secondary to a major physical condition (consultation will be sought from medical professionals where appropriate on an individual basis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Anxiety and/or depression in Type 2 Diabetes | 18 weeks
  To see whether a CBT based guided self-help book improves anxiety and/or depression in participants with Type 2 Diabetes

SECONDARY OUTCOMES:
Quality of life | 18 weeks
  To see whether the intervention enhances quality of life, psychological well-being and self-reported diabetes management.

CONTACTS AND LOCATIONS:
Locations (1):
- Raigmore Hospital, Inverness, Highlands, United Kingdom